CLINICAL TRIAL: NCT05414435
Title: Informed Consent in Endoscopy: Read, Understood or Merely Signed?
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar Tondela-Viseu (Other)
Responsible Party: Principal Investigator, Ana Carvalho, Principal Investigator, Centro Hospitalar Tondela-Viseu
Other Study IDs: CHTV07/2022.1
Record Dates: First submitted 2022-06-05; First posted 2022-06-10 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Informed Consent; Gastrointestinal Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Reading of informed consent form — Patients that adequately read informed consent forms

SUMMARY:
Informed consent form is a legal document that, ethically, should be obtained before any endoscopic procedure is performed.

The main purpose of this research study is to assess the readability, comprehensibility and applicability of the new informed consent proposed by the Portuguese Society of Digestive Endoscopy as a way to standardize the information provided to patients prior to endoscopic exams.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients able to autonomously give informed consent
* Patients refered to elective endoscopic procedures (upper digestive endoscopy and/or colonoscopy) without deep sedation.

Exclusion Criteria:

* Patients refered to urgent endoscopic procedures
* Patients refered for endoscopic procedures with deep sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients refered for elective endoscopic procedures
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Assessing the percentage of patients who adequate read informed consent forms | 12 months
  Assess if patients "adequately read" informed consent forms - "adequate reading" was defined by checking all of the following: signing of informed consent form; fulfilment of a questionnaire regarding medical history and drugs; underlining a small sentence added to the orignial version of informed consent form.
  Patients not meeting all the defined criteria were considered not to have adequately read the informed consent.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Cardoso, MD, Study Director — Centro Hospitalar Tondela-Viseu, E.P.E.
Locations (1):
- Centro Hospitalar Tondela Viseu, Viseu, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carvalho AC, Cardoso R, Vieira HM, Silva A. Informed consent in endoscopy: Read, understood, or just signed? IGIE. 2024 Apr 9;3(2):222-229. doi: 10.1016/j.igie.2024.04.001. eCollection 2024 Jun. PMID 41647094